CLINICAL TRIAL: NCT00289276
Title: FAST (Fluid Accumulation Status Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: CRDM Clinical, Medtronic CRDM
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 228
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Congestive Heart Failure; Cardiomyopathy; Dyspnea; Pulmonary Edema; Heart Diseases
Keywords: Cardiomyopathy; Ventricular Ejection Fraction; Congestive Heart Failure; Impedance
MeSH Terms: conditions — Heart Failure; Cardiomyopathies; Dyspnea; Pulmonary Edema; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fluid Status Monitoring (OptiVol™) — Thoracic Fluid Status Software downloaded on all subjects enrolled in the trial

SUMMARY:
Heart failure is a progressive disease that decreases the pumping action of the heart. This may cause a backup of fluid in the heart and may result in heart beat changes. Using very low electrical pulses that travel across the inside of the chest cavity, thoracic fluid status monitoring (OptiVol™) can measure the level of resistance to the electrical pulses, which indicates the level of fluid in the chest. The purpose of this study is to collect information related to fluid build up in the chest of subjects with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with one of the following implantable cardioverter defibrillators (ICDs): InSync Marquis™, InSync II Marquis™, Marquis® DR, or InSync III Marquis™.
* Subjects with an ICD placed in the upper part of the left or right side of their chest.
* Subjects with a lead (flexible wire that sends electrical signals from the ICD directly to the heart tissue) that is inserted through a vein and placed in the right ventricle (RV) of the heart (a transvenous RV lead).
* Subjects who underwent the ICD implant procedure, or any readjusting of the ICD, 30 days or more prior to enrolling in the study.

Exclusion Criteria:

* Subjects who are already enrolled in another clinical study.
* Subjects who have received a heart transplant.
* Subjects who are unable or unwilling to follow the study schedule of visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2003-11; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (12):
  - Alaska Cardiovascular Research Foundation, Anchorage, Alaska
  - Palm Beach Heart Institute, Atlantis, Florida
  - Fort Wayne Cardiology, Fort Wayne, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - North Shore University Hospital, Manhasset, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation Department of Hear Failure/Transplantation, Cleveland, Ohio
  - The Ohio State University Hospital, Columbus, Ohio
  - The Pavillion at Doylestown Hospital, Doylestown, Pennsylvania
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Intermountain Medical Center, Salt Lake City, Utah
- Canada (2):
  - University of Calgary/Foothills Hospital, Calgary, Alberta
  - Kingston General Hospital, Kingston, Ontario
- China (2):
  - Queen Mary Hospital, Pok Fu Lam, Hong Kong
  - Prince of Wales Hospital/The Chinese University of Hong Kong, Shatin, Hong Kong

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were two parts to the FAST study. The first part was called FAST Pivotal and the second part was called FAST Expansion. Subjects were enrolled in the FAST study from November 2003 through September 2007. Subject follow-ups were complete and all subjects were exited by April 2008.
Pre-assignment Details: None of the subjects in FAST Pivotal were included in FAST Expansion.
Groups:
- FAST Pivotal: FAST Pivotal was the first part of the FAST study. Subjects were enrolled under the Clinical Investigation Plan (CIP) Versions 2.0/3.0 from November 2003 to November 2004. The purpose of this part of the FAST study was to collect intra-thoracic impedance data required to support the approval of the Fluid Status Trend feature.
- FAST Expansion: FAST Expansion is the second part of the FAST study. Subjects were enrolled under the CIP Versions 7.0/8.0 and 10/11 from January 2005 to September 2007. The purpose of this part of the FAST study was to expand on the FAST Pivotal study by collecting additional intra-thoracic impedance data to gain more experience with the Fluid Status Trend feature.
Period: First Part of FAST Study (Pivotal)
Arm/Group | FAST Pivotal | FAST Expansion
Started | 47 (11 patients were re-consented under version 7 of the CIP, but are included in Pivotal results only) | 0
Completed | 47 | 0
Not Completed | 0 | 0
Period: Second Part of FAST Study (Expansion)
Arm/Group | FAST Pivotal | FAST Expansion
Started | 0 | 109
Completed | 0 | 106
Not Completed | 0 | 3
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FAST Pivotal | FAST Expansion | Total
Number analyzed (Participants) | 47 | 109 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 15 | 29 | 44.0
  >=65 years | 32 | 80 | 112.0
Age Continuous [Mean (Standard Deviation); unit: years] | 68.8 (10.5) | 69.6 (11.1) | 69.4 (10.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 26 | 36.0
  Male | 37 | 83 | 120.0
Region of Enrollment [Number; unit: participants]
  United States | 41 | 90 | 131.0
  Canada | 6 | 5 | 11.0
  China | 0 | 14 | 14.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least 30 Days of Daily Impedance Measurements
Description: Impedance measurements were presented graphically over time in relation to clinical events for all subjects with at least 30 days of follow-up and impedance data collected during the follow-up period.
Time Frame: Up to 36 months.
Population: Includes all enrolled participants.
Measure: Number; unit: participants
Arm/Group | FAST Pivotal | FAST Expansion
Number analyzed (Participants) | 47 | 109
participants | 47 | 106

2. Secondary Outcome: Change in Thoracic Impedance Associated With Heart Failure (HF) Hospitalization for an Exacerbation of HF
Description: Difference in mean thoracic impedance: post-hospitalization minus pre-hospitalization.
Time Frame: 3 days pre-admission and 3 days post-discharge
Population: All subjects with at least one heart failure hospitalization and with impedance data pre and post-hospitalization.
Measure: Mean (Full Range); unit: Ohms
Arm/Group | FAST Pivotal | FAST Expansion
Number analyzed (Participants) | 5 | 23
Ohms | 2.50 [-7.50 to 10.58] | 2.93 [-17.17 to 11.08]

3. Secondary Outcome: Change in Thoracic Impedance Associated With Heart Failure (HF) Outpatient Treatment of an Exacerbation of HF
Description: Difference in mean thoracic impedance: post-outpatient visit minus pre-outpatient visit.
Time Frame: 1 day pre and 1 day post-outpatient visit
Population: All subjects with at least one heart failure outpatient treatment and with impedance data pre and post-outpatient treatment.
Measure: Mean (Full Range); unit: Ohms
Arm/Group | FAST Pivotal | FAST Expansion
Number analyzed (Participants) | 1 | 4
Ohms | 6.00 [6.00 to 6.00] | 0.00 [-4.50 to 7.00]

4. Secondary Outcome: Number of Adverse Events
Description: All adverse events were collected for this trial such as (but not limited to): Atrial Fibrillation, Chest Pain, Pneumonia, Cold/Flu
Time Frame: From enrollment to study exit (up to 36 months).
Population: Number of participants analyzed for this outcome is limited to subjects who experienced at least one Adverse Event from enrollment to study exit.
Measure: Number; unit: Adverse Events
Arm/Group | FAST Pivotal | FAST Expansion
Number analyzed (Participants) | 41 | 94
Adverse Events | 154 | 421

ADVERSE EVENTS:
Time Frame: From enrollment to study exit (up to 36 months).
Description: For this study a serious adverse event was defined as an adverse event which results in invasive treatment or which directly results in the death or serious injury to the subject, or the termination of significant device function regardless of other treatments.
Arm/Group | FAST Pivotal | FAST Expansion
Serious Adverse Events (participants affected / at risk) | 33/47 | 76/109
Other Adverse Events (participants affected / at risk) | 20/47 | 52/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAST Pivotal (N=47) | FAST Expansion (N=109)
Arm/Hand Swelling (General disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (General disorders) | 0 (0) | 5 (5)
Back Pain/Discomfort (General disorders) | 0 (0) | 1 (1)
Cancer (General disorders) | 2 (2) | 1 (1)
Cardiomyopathy (General disorders) | 0 (0) | 3 (3)
Chest Pain/Angina Pectoris (General disorders) | 1 (1) | 6 (6)
Chest Pressure/Tightness (General disorders) | 1 (1) | 1 (1)
Chronic Obstructive Pulmonary Disease (General disorders) | 0 (0) | 2 (2)
Cold/Flu (General disorders) | 0 (0) | 1 (1)
Dehydration (General disorders) | 1 (1) | 1 (1)
Diabetes (General disorders) | 0 (0) | 2 (2)
Fatigue/Tiredness (General disorders) | 1 (1) | 1 (1)
Heart Failure Decompensation (General disorders) | 10 (16) | 28 (63)
Hypokalemia (General disorders) | 0 (0) | 1 (1)
Hypotension (General disorders) | 0 (0) | 3 (3)
Ischemic Heart Disease (General disorders) | 0 (0) | 1 (1)
Lead Conductor Fracture (General disorders) | 0 (0) | 1 (1)
Lead Dislodgment (General disorders) | 0 (0) | 1 (1)
Muscle Stimulation - Diaphragm (General disorders) | 1 (1) | 1 (1)
Myocardial Infarction (General disorders) | 1 (1) | 2 (2)
Other: Aberrantly Conducted Rhythm (General disorders) | 0 (0) | 1 (1)
Other: Acute Cystitis (General disorders) | 1 (1) | 0 (0)
Other: Amiodarone Toxicity (General disorders) | 0 (0) | 1 (1)
Other: Anemia (General disorders) | 1 (1) | 1 (3)
Other: Arm Pain (General disorders) | 0 (0) | 1 (1)
Other: Battery at Elective Replacement Indicator (General disorders) | 3 (3) | 29 (29)
Other: COAG - Negative Staphylococcus Bacteremia (General disorders) | 1 (1) | 0 (0)
Other: Cardiac Arrest (General disorders) | 0 (0) | 1 (1)
Other: Cataracts (General disorders) | 0 (0) | 2 (2)
Other: Cholecystitis (General disorders) | 0 (0) | 1 (1)
Other: Clostidium Difficile Colitis Infection (General disorders) | 0 (0) | 1 (1)
Other: Cushing's Syndrome (General disorders) | 0 (0) | 1 (1)
Other: Diverticular Disease (General disorders) | 1 (1) | 0 (0)
Other: Effusion of Right Knee Joint (General disorders) | 0 (0) | 1 (1)
Other: Enlarged Prostate (General disorders) | 0 (0) | 1 (1)
Other: Epicardial Lead Placement in Lateral Wall-Poor Placement (General disorders) | 0 (0) | 1 (1)
Other: Fall (General disorders) | 0 (0) | 2 (2)
Other: Fractured Femur (General disorders) | 1 (1) | 0 (0)
Other: Gastrointestinal Bleed (General disorders) | 0 (0) | 2 (2)
Other: Head Injury (General disorders) | 0 (0) | 1 (1)
Other: High INR (General disorders) | 0 (0) | 1 (1)
Other: Inappropriate Shock (General disorders) | 0 (0) | 1 (1)
Other: Indigestion (General disorders) | 1 (1) | 0 (0)
Other: Infected Carbuncle (General disorders) | 0 (0) | 1 (1)
Other: Infected Fistula (gortex) Right Arm (General disorders) | 1 (1) | 0 (0)
Other: Infected Sebaceous Cyst (General disorders) | 0 (0) | 1 (1)
Other: Infection (General disorders) | 0 (0) | 1 (1)
Other: Inguinal Hernia (General disorders) | 0 (0) | 1 (1)
Other: Iron Deficiency Anemia / GI Bleed (General disorders) | 0 (0) | 1 (1)
Other: Kidney Stones (General disorders) | 0 (0) | 1 (1)
Other: Left Indirect Inguinal Hernia (General disorders) | 0 (0) | 1 (1)
Other: Leg Cramps (General disorders) | 0 (0) | 1 (1)
Other: Marquis Battery Field Action (General disorders) | 14 (14) | 5 (5)
Other: Melena (General disorders) | 0 (0) | 1 (1)
Other: Non-functioning Fistula (General disorders) | 1 (1) | 0 (0)
Other: Osteoarthritis (General disorders) | 0 (0) | 1 (1)
Other: Pain/Swelling Elbows Bilaterally (General disorders) | 0 (0) | 1 (1)
Other: Pancreatitis (General disorders) | 0 (0) | 1 (1)
Other: Peptic Ulcers (General disorders) | 0 (0) | 1 (1)
Other: Poorly Functioning Fistula (General disorders) | 1 (3) | 0 (0)
Other: Prostate Enlargement (General disorders) | 0 (0) | 1 (1)
Other: Prostate Problems (General disorders) | 0 (0) | 1 (1)
Other: Renal Colic (General disorders) | 0 (0) | 1 (1)
Other: Right Carotid Artery Stenosis (General disorders) | 1 (1) | 0 (0)
Other: SVT-Classified as VT with Therapies Delivered (General disorders) | 0 (0) | 1 (1)
Other: Sepsis (General disorders) | 0 (0) | 1 (1)
Other: Sepsis Syndrome (General disorders) | 0 (0) | 1 (1)
Other: Severe Anemia (General disorders) | 1 (1) | 1 (1)
Other: Small Bowel Malformation (General disorders) | 1 (1) | 0 (0)
Other: Small Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other: Stenosis of the Transposed Vessilic Vein (General disorders) | 1 (1) | 0 (0)
Other: Subclavian Artery Stenosis (General disorders) | 0 (0) | 1 (1)
Other: Urinary Tract Infection (General disorders) | 0 (0) | 3 (3)
Other: Uterine Ablation (General disorders) | 1 (1) | 0 (0)
Other: Weight Loss, Night Sweats, Chills (General disorders) | 0 (0) | 1 (1)
Other: Worsening Osteoarthritis (General disorders) | 0 (0) | 1 (1)
Oversensing (General disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disease (General disorders) | 1 (1) | 1 (1)
Pneumonia (General disorders) | 1 (1) | 6 (8)
Premature Battery Failure (General disorders) | 5 (5) | 0 (0)
Rash (General disorders) | 0 (0) | 1 (1)
Renal Failure (General disorders) | 2 (2) | 10 (10)
Stroke/CVA (General disorders) | 1 (1) | 1 (1)
Suspected Generator/ICD Failure (General disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 0 (0) | 1 (1)
Thrombosis (General disorders) | 0 (0) | 1 (1)
Ventricular Tachycardia (General disorders) | 0 (0) | 2 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAST Pivotal (N=47) | FAST Expansion (N=109)
Bronchitis (General disorders) | 0 (0) | 6 (6)
Chest Pain/Angina Pectoris (General disorders) | 0 (0) | 8 (8)
Cold/Flu (General disorders) | 5 (5) | 14 (16)
Dizziness (General disorders) | 6 (6) | 6 (7)
Dyspnea/Shortness of Breath (General disorders) | 4 (4) | 8 (8)
Fatigue/Tiredness (General disorders) | 4 (4) | 0 (0)
Heart Failure Decompensation (General disorders) | 4 (4) | 11 (13)
Other: Battery at Elective Replacement Indicator (General disorders) | 0 (0) | 7 (7)
Other: Fall (General disorders) | 3 (4) | 0 (0)
Ventricular Tachycardia (General disorders) | 3 (3) | 9 (14)

LIMITATIONS AND CAVEATS:
This was a characterization study with no descriptive statistical analysis. The results reported were counts of subjects with impedance data available as applicable for each objective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, contracts allow investigators ("PI") to publish per the publication strategy/Clinical Investigation Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), and (b) selection and order of publications by the publications committee. Any such CI is deleted prior to publication/presentation. Medtronic may not otherwise censor/interfere with the publication. PI's may not publish single-site data until the main multi-site publication has occurred.